CLINICAL TRIAL: NCT00044629
Title: Combined Behavioral/Pharmacological Therapy for Insomnia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00011850; R01MH062119 (NIH); DSIR 83-ATAS
Record Dates: First submitted 2002-09-03; First posted 2002-09-05 (Estimated); Last update posted 2013-09-16 (Estimated); Status verified 2013-09

CONDITIONS: Sleep Initiation and Maintenance Disorders
Keywords: Sleep Deprivation; Insomnia; Sleep Disorders
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Sleep Deprivation; Sleep Wake Disorders | interventions — Cognitive Behavioral Therapy; Zolpidem

ARMS (3):
- Cognitive Behavioral Therapy and Ambien (Experimental): Cognitive Behavioral Therapy and Ambien
  Interventions: Behavioral: Cognitive-Behavioral Therapy for Insomnia; Drug: zolpidem tartrate (Ambien)
- Cognitive Behavioral Therapy and Placebo (Placebo Comparator): Cognitive Behavioral Therapy and Placebo
  Interventions: Behavioral: Cognitive-Behavioral Therapy for Insomnia; Drug: Placebo
- Cognitive Behavioral Therapy alone (no drug) (Active Comparator): Cognitive Behavioral Therapy alone (no drug)
  Interventions: Behavioral: Cognitive-Behavioral Therapy for Insomnia

INTERVENTIONS:
Behavioral: Cognitive-Behavioral Therapy for Insomnia
Drug: zolpidem tartrate (Ambien)
  Arms: Cognitive Behavioral Therapy and Ambien
Drug: Placebo
  Arms: Cognitive Behavioral Therapy and Placebo

SUMMARY:
This study will determine how sleeping pills can be combined with nondrug treatments to maximize the benefits of therapy for insomnia.

DETAILED DESCRIPTION:
Long-term insomnia is a common and significant health problem. Two main treatments, pharmacotherapy and behavioral therapy, have been used to help people with insomnia. Because both treatments have advantages and disadvantages, a combination of these treatments may be a good way to treat insomnia.

During the first 2 weeks of the study, participants keep a sleep log, wear an actigraph (a device that resembles a wristwatch and records activity to help determine when participants are asleep or awake), and complete questionnaires.

Participants are then randomly assigned to receive 6 weeks of behavioral therapy plus zolpidem tartrate (Ambien), behavioral therapy plus placebo, or behavioral therapy alone. During treatment, participants return to the clinic once a week to turn in their sleep logs, download their actigraph, and complete questionnaires.

After 6 weeks, participants enter the post-treatment phase of the study, which lasts 2 weeks and is identical to the 2-week assessment at the beginning of the study.

After the post-treatment phase, participants enter the follow-up period and are contacted at 3 months, 6 months, and 1 year to complete another 2-week assessment with sleep logs, actigraphy, and questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* be between 21 and 75 years of age
* have a mean total nocturnal wake time of > 60 min./night
* have a history of insomnia > 6 months
* have a history of one or more poor sleep hygiene practices such as taking 3 or more naps/week, varying bed times or wake times by > 2 hrs. from day to day, or routinely lying in bed awake for periods > 30 min

Exclusion Criteria:

* pregnant women
* the terminally ill
* individuals with other medical conditions (e.g. chronic pain disorders, etc.) that compromise sleep
* individuals with major psychiatric diagnoses
* persons with hypnotic-dependent insomnia
* subjects on antidepressants or anxiolytics
* subjects with evidence of sleep apnea

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2001-09; Study Completion 2006-08

CONTACTS AND LOCATIONS:
Locations (1):
- Duke Sleep Disorders Center, Durham, North Carolina, United States